CLINICAL TRIAL: NCT03710746
Title: Enhancing Effectiveness of a Dissonance-Based Obesity Prevention Program
Brief Title: Project Health: Enhancing Effectiveness of a Dissonance-Based Obesity Prevention Program
Acronym: PH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HD093598-01A1
Record Dates: First submitted 2018-10-08; First posted 2018-10-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight; prevention; adolescence; dissonance
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to their response training condition. Outcomes assessors will be masked to both participant conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Mixed Group, Food Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in mixed-sex groups and will complete the food-focused response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Mixed Group, Generic Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in mixed-sex groups and will complete the generic response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Female Group, Food Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in female-only groups and will complete the food-focused response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Female Group, Generic Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in female-only groups and will complete the generic response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Male Group, Food Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in male-only groups and will complete the food-focused response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training
- Male Group, Generic Response Training (Experimental): Participants in this arm will be assigned to receive Project Health in male-only groups and will complete the generic response and attention training intervention.
  Interventions: Behavioral: Project Health; Behavioral: Response and Attention Training

INTERVENTIONS:
Behavioral: Project Health — A brief dissonance-based obesity prevention program delivered in six one-hour weekly sessions.
Behavioral: Response and Attention Training — Individualized, computerized response and attention training consisting of five separate tasks designed to increase inhibitory control to reduce overeating.

SUMMARY:
This project seeks to improve the effectiveness of a novel dissonance-based obesity prevention program that has reduced future BMI gain and overweight/obesity onset by (a) experimentally testing whether implementing it in single- versus mixed-sex groups, which should increase dissonance-induction that contributes to weight gain prevention effects, and (b) experimentally testing whether adding food response and attention training, which theoretically reduces valuation of and attention for high-calorie foods, increases weight gain prevention effects. This randomized trial would be the first to experimentally manipulate these two factors in an effort to produce superior weight gain prevention effects. A brief effective obesity prevention program that can be easily, inexpensively, and broadly implemented to late adolescents at risk for excess weight gain, as has been the case with another dissonance-based prevention program, could markedly reduce the prevalence of obesity and associated morbidity and mortality.

DETAILED DESCRIPTION:
Prevention is key for combating obesity, but few programs have prevented future increases in BMI and onset of overweight/obesity, particularly during late adolescence when youth often assume responsibility for dietary intake and exercise choices. One exception is a brief 6-hr dissonance-based program (Project Health) wherein participants make small lasting incremental lifestyle changes to dietary intake and exercise to reach energy balance, and discuss costs of obesity, an unhealthy diet, and sedentary behavior, and benefits of leanness, a healthy diet, and exercise, which prompts them to align their attitudes with their publicly displayed behavior. These activities promote the internalization of health goals and executive control over lifestyle behaviors. Late adolescents randomized to Project Health showed fewer increases in BMI and a 41% and 43% reduction in overweight/obesity onset over 2-yr follow-up compared to a version of the program lacking dissonance induction activities and an obesity education condition. Project Health appears to be the first program to produce these key obesity prevention effects relative to an alternative intervention, but it is critical to increase effects. A dissonance-based prevention program was more effective when implemented in single- versus mixed-sex groups, theoretically, because it promoted greater participation in dissonance-inducing discussions. Aim 1a is to test whether the weight gain prevention effects will be larger when Project Health is implemented in single-sex groups; the investigators will randomize 450 17-20-year-olds to complete Project Health in female, male, or mixed-sex groups, assessing outcomes at pretest, post-test, and 6, 12, 24, and 36-month follow-ups. Aim 1b is to test whether greater participation in dissonance-inducing discussions and group cohesion mediate the effect of condition on any superior weight gain prevention effects. Adolescents who show greater functional Magnetic Resonance Imaging( fMRI)-assessed reward and attention region responsivity to food images exhibit elevated future weight gain, implying that reducing this responsivity may reduce future weight gain. In a pilot trial, late adolescents who completed go/no-go, stop-signal, and respond-signal computer training in which they repeatedly inhibit responses to high-calorie foods and respond to low-calorie foods, and dot-probe and visual-search computer tasks that train attention away from high-calorie foods and to low-calorie foods, showed a greater reduction in reward and attention region responsivity to, palatability rating of, and willingness to pay for, high-calorie foods, suggesting reduced valuation and attentional bias, as well as greater fat loss over 1-yr follow-up versus controls who completed the training with non-food images. Aim 2a is to test whether adding food response and attention training to Project Health will produce larger weight gain prevention effects. Participants in the 3 conditions will be randomized to complete response and attention training for 25-mins after each of the 6-sessions with either food or non-food images. Aim 2b is to test whether reduced palatability ratings of, willingness to pay, and attentional bias for high-calorie foods mediate the effect of training condition on any superior weight gain prevention effects.

During the Coronavirus Disease 2019 (COVID-19) shelter-at-home order, the investigators will not measure in-person only outcomes including assessments using the BodPod (a body composition tracking system using air displacement plethysmography), and height and weight measurement for BMI calculation for all participants that have assessments due during this order. The investigators will continue to conduct intervention groups that will be administered on a virtual platform.

ELIGIBILITY:
Inclusion Criteria:

* Current at least moderate weight concerns (response of moderate, severe or extreme to the presence of weight concerns question)
* BMI between 20 and 30

Exclusion Criteria:

* Current diagnosis of anorexia nervosa, bulimia nervosa, or binge eating disorder

Ages: 17 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 406 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Body Fat | Baseline, 2 months, 8 months, 14 months, 26 months, and 38 months
  Change in percentage of body fat (Not collected during COVID-19 shelter-at-home order)

SECONDARY OUTCOMES:
Weight Concerns Scale from the Eating Disorder Examination Questionnaire (EDE-Q) | Baseline, 2 months, 8 months, 14 months, 26 months, and 38 months
  Change in weight concerns. Scale scores range from 0 to 42 with higher scores being indicative of higher weight concerns.
Beck Depression Index (BDI) | Baseline, 2 months, 8 months, 14 months, 26 months, and 38 months
  Change in depressive symptoms
Eating Disorder Interview (EDDI) | Baseline, 2 months, 8 months, 14 months, 26 months, and 38 months
  Change in eating disorder symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Stice, Ph.D., Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - Oregon Research Institute, Eugene, Oregon
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share all study data via the NICHD Data and Specimen Hub (DASH), which is the centralized resource for researchers to store and access data from NICHD-funded research studies to use for secondary research. All data, with the exception of video recordings of the participants in treatment (which cannot be effectively de-identified), will be provided.
Time Frame: After all follow-up assessments are completed and the main project papers are published, a dataset stripped of identifiers prior to release will be made available without cost to researchers and analysts.
Access Criteria: Individuals wishing to view Individual Participant Data (IPD) can create a free user account at DASH and submit a request which will be reviewed and approved through the NICHD Dash administrator.

REFERENCES:
- See also: Oregon Research Institute Website — http://www.ori.org
- See also: Drexel University: WELL Center Website — http://drexel.edu/coas/academics/departments-centers/well-center/